CLINICAL TRIAL: NCT00777010
Title: Energy Metabolism and Cognitive Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Robert Krikorian, Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 04-09-17-01
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Mild Cognitive Impairment
Keywords: memory loss; mild cognitive impairment; forgetfulness
MeSH Terms: conditions — Cognitive Dysfunction; Memory Disorders | interventions — Diet, Ketogenic

STUDY DESIGN:
Intervention Model Description: Parallel groups, randomized controlled nutritional intervention.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy high carbohydrate diet (Active Comparator): Participants will follow a typical, higher carbohydrate dietary intervention with emphasis on lower glycemic carbohydrate foods and monounsaturated fatty acid consumption
  Interventions: Other: Healthy high carbohydrate diet
- Carbohydrate restricted, ketogenic diet (Experimental): Paricipants will follow a carbohydrate restricted dietary intervention designed to induce ketone metabolism
  Interventions: Other: Ketogenic diet

INTERVENTIONS:
Other: Ketogenic diet — carbohydrate restricted diet
  Arms: Carbohydrate restricted, ketogenic diet
Other: Healthy high carbohydrate diet — higher carbohydrate diet
  Arms: Healthy high carbohydrate diet

SUMMARY:
Participants 60 and older with and without Parkinson's disease who have mild cognitive decline will be randomized to either a standard higher carbohydrate diet or a carbohydrate-restricted ketogenic diet for 8 weeks. The main hypothesis is that nutritional ketosis will improve memory functioning. Pre and post-memory testing will be performed. Subjects will also provide blood samples and a subset of subjects with receive magnetic resonance brain imaging.

DETAILED DESCRIPTION:
Obesity and metabolic disturbance are recognized as important risks for disorders such as cardiovascular disease, stroke, and cancer. However, these conditions also contribute to age-related cognitive decline and dementia. In particular, insulin resistance and hyperinsulinemia promote neurocognitive dysfunction and neurodegenerative changes during the extended pre-clinical phase of Alzheimer's disease (AD). The prevalence of both metabolic disturbance and dementia are increasing dramatically, and in the absence of effective treatment, preventive approaches are essential to address the ominous public health concern represented by Alzheimer's disease and other forms of dementia. Dietary intervention is a promising and under-investigated preventive option. Regimens involving restricted carbohydrate consumption designed to induce ketone metabolism have been shown to improve metabolic parameters. In addition, ketone metabolism is associated with a host of benefits for neural function, among them enhanced mitochondrial energy production and reduction of neuropathological factors. Ketone feeding studies have demonstrated acute functional improvement in older adults with neurocognitive decline.

This research is designed to assess the efficacy of strict carbohydrate restriction in correcting hyperinsulinemia and improving neurocognitive function in older adults with early memory decline. Recently, we have shown that relatively brief intervention involving a low carbohydrate, ketogenic diet can improve memory in subjects with Mild Cognitive Impairment. We would like to extend these initial findings by adding new study arms involving older adult subjects with Parkinson's disease and Mild Cognitive Impairment. We also will increase the intervention period from six weeks to eight weeks.

Aim 1: To evaluate the effect of adaptation to ketosis on cognitive function in older adults with Age-Associated Memory Impairment (AAMI) and Mild Cognitive Impairment (MCI).

Hypothesis 1. Subjects with AAMI and MCI will show improved working memory and long-term memory ability after practicing a low carbohydrate, ketogenic diet for six weeks relative to comparison subjects who maintain a typical, high carbohydrate, nonketogenic diet.

Aim 2: To assess the effect of ketone metabolism on memory and motor function in subjects with Parkinson's disease and Mild Cognitive Impairment after eight (8) weeks of dietary intervention.

Hypothesis 2. Subjects with Parkinson's disease and MCI will show improved working memory and long-term memory function after practicing a low carbohydrate, ketogenic diet for eight weeks relative to comparison subjects who consume a typical, high carbohydrate nonketogenic diet.

Hypothesis 3. Subjects with Parkinson's disease and MCI will show improved motor function after practicing a low carbohydrate, ketogenic diet for eight weeks relative to comparison subjects who consume a typical, high carbohydrate nonketogenic diet.

We also will evaluate changes in mood, ketone body levels, serum lipids, inflammatory markers, and fasting glucose and insulin and assess relationships of these factors with the primary outcome measures. We will obtain diet records during the intervention to assess adherence to the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years or older
* Mild cognitive impairment

Exclusion Criteria:

* Diabetes
* Medications that have effect on memory
* Memory problems due to medical issues (ie head injury, stroke, untreated sleep apnea etc.)
* Unable to complete an MRI scan

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2008-09-01; Primary Completion 2016-12-31 (Actual); Study Completion 2017-03-15 (Actual)

PRIMARY OUTCOMES:
improvement in memory testing | 6 or 8 weeks

SECONDARY OUTCOMES:
correlation between diet, metabolic factors, memory performance, and cerebral activation | 6 or 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert Krikorian, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No